CLINICAL TRIAL: NCT05197569
Title: The Effect of Aromatherapy With Thyme Oil on Disease Symptoms, Vital Signs and Hemodynamic Parameters in COVID-19 Patients
Brief Title: The Effect of Aromatherapy With Thyme Oil on Disease Symptoms, Vital Signs, Hemodynamic Parameters in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/2637
Record Dates: First submitted 2022-01-03; First posted 2022-01-19 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Patient Engagement
Keywords: Coronavirus; Covid-19; Aromatherapy; thyme oil; Thymus vulgaris
MeSH Terms: conditions — Patient Participation; Coronavirus Infections; COVID-19 | interventions — thyme oil

STUDY DESIGN:
Intervention Model Description: In the study, patients will be stratified according to their gender (male and female) status and the blocking process will be performed. In this study, block randomization will be done according to age groups in order to assign the participants to the experimental and control groups. Patients will be listed according to the hospitalization list and numbered up to 140. Numbers will be assigned to the experimental and control groups according to the random numbers list. Thus, the probability of each patient in the groups being in either of the intervention or control groups will be equalized.
  Group 1: experimental 2. Group: Control
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention will be applied to the control group and the measurements will be recorded simultaneously.
- Thyme oil group (Experimental): After filling out the forms, thyme oil aromatherapy will be applied to the patients assigned to the experimental group .The oregano oil to be prepared must have a high carvacrol ratio. Thyme oil with a carvacrol ratio of at least 74% will be specific to each patient and will be given to the patient in the form of an inhaler stick. According to expert opinion; The patient's own room should be visited every 8 hours and the patient-specific inhaler stick should be sniffed into 8 breathing lungs. Each patient will use an inhaler stick for 5 days. Hemodynamic parameters (ph, CO 2, O 2 ) and Covid-19 symptoms will be measured before the intervention with the patient (pretest) and at the end of the 5th day (posttest). Vital signs will be measured and recorded three times a day in the patient's room at 08:00, 16:00 and 24:00.
  Interventions: Other: thyme oil

INTERVENTIONS:
Other: thyme oil — Thyme oil with a carvacrol ratio of at least 74% will be specific to each patient and will be given to the patient in the form of an inhaler stick. According to expert opinion; The patient's own room should be visited every 8 hours and the patient-specific inhaler stick should be sniffed into 8 breathing lungs. Each patient will use an inhaler stick for 5 days. Hemodynamic parameters (ph, CO 2, O 2 ) and Covid-19 symptoms will be measured before the intervention with the patient (pretest) and at the end of the 5th day (posttest). Vital signs will be measured and recorded three times a day in the patient's room at 08:00, 16:00 and 24:00.
  Arms: Thyme oil group

SUMMARY:
Coronavirus, which is a common infectious disease, is characterized by symptoms such as severe pain, cough, shortness of breath, dizziness, secretion, diarrhea, nausea-vomiting, weakness, runny nose, changes in sense of taste and smell, and loss of appetite. The use of thyme is common for this disease whose standard treatment is still being discussed. However, studies investigating the effectiveness of oregano oil are limited. These few studies in the literature have focused especially on the effects of thyme oil on Covid-19 symptoms. This work; It will be done to evaluate the effect of aromatherapy with thyme oil on Covid-19 symptoms, vital signs and hemodynamic parameters in Covid-19 patients. There is no study in the literature investigating the effects of all these variables.

DETAILED DESCRIPTION:
Coronavirus, which is a common infectious disease, is characterized by symptoms such as severe pain, cough, shortness of breath, dizziness, secretion, diarrhea, nausea-vomiting, weakness, runny nose, changes in sense of taste and smell, and loss of appetite. The use of thyme is common for this disease whose standard treatment is still being discussed. However, studies investigating the effectiveness of oregano oil are limited. These few studies in the literature have focused especially on the effects of thyme oil on Covid-19 symptoms. This work; It will be done to evaluate the effect of aromatherapy with thyme oil on Covid-19 symptoms, vital signs and hemodynamic parameters in Covid-19 patients. There is no study in the literature investigating the effects of all these variables. The study will be carried out as a randomized controlled experimental study. It will be carried out in Batman Training and Research Hospital Covid-19 service between January 2022 and December 2022. The sample of the study will consist of a total of 140 patients (experimental group = 70 control group = 70) randomized to the experimental and control groups.

In data collection, "Demographic Characteristics Form", "Covid-19 Symptom Form", "Hemodynamic parameters and vital signs follow-up form" and "Visual Comparison Scale (VAS)" will be used. Kolmogorov Smirnov normality test will be used for normal distribution in the analysis of the data. Using ANOVA, ANCOVA, student t test and paired t test in the analysis of normally distributed data; Fridman test, Kruskal Wallis and Man Withney U test are planned to be used in the analysis of data that is not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* PCR test positive
* Being in the covid-19 service
* Involvement in the lung as a result of computed tomography between 50-80% to be
* The day of admission to the Covid 19 service (1. Day) sickareceipt of

Exclusion Criteria:

* Having a pregnancy status
* be under the age of 18
* unwillingness to participate in the study
* Patients who will be transferred to the intensive care unit will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Demographic Characteristics Form | 6 months
  This form, created by the researchers, consists of 10 questions in total, questioning the characteristics of diagnosis, weight, gender, chronic disease status and Covid-19 .
Covid-19 Symptom Form | 6 months
  This form, which was created by the researchers with the support of the literature, consists of 13 questions that include evaluations that measure the patient's Covid-19 symptoms and the level of severity.
Hemodynamic parameters form | 6 months
  From the blood gas values of this form created by the researcher; It was created to record the pH, O 2 , CO 2 , SaO 2 measurement results.
Visual Comparison Scale | 6 months
  This scale is the most widely used scale for pain assessment. In this study, it will be used for the evaluation of muscle-joint pain and headache, which are the symptoms of Covid-19. Usually 10 cm long, horizontally or vertically; It is the line from "No Pain" (0 point) to "Severe Pain" (10 points). As the score on the visual comparison scale increases, the severity of the disease increases. This line can be straight or vertical. It may include words or numbers used to describe pain, written on evenly spaced lines. It is generally accepted that the horizontal line is easier to understand.
Vital signs follow-up form | 6 months
  Vital signs follow-up form was created to record the patient's daily fever, pulse, respiratory rate, systolic diastolic blood pressure values.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Training and Research Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This research is a doctoral thesis study. The research is expected to be completed.